CLINICAL TRIAL: NCT01666262
Title: Phase I/II Safety and Immunogenicity of Pandemic Live Attenuated Influenza Vaccine (PLAIV) Candidate Strain A/17/CA/2009/38 (H1N1) in Healthy Thais
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GPO FLU VACCINE-01
Record Dates: First submitted 2010-01-11; First posted 2012-08-16 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: FLU; H1N1; GPO; PLAIV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A/17/CA/2009/38 (H1N1) (Experimental)
  Interventions: Biological: Vaccine A/17/CA/2009/38 (H1N1)
- Stabilizer (Placebo Comparator)
  Interventions: Other: Placebo:Stabilizer

INTERVENTIONS:
Biological: Vaccine A/17/CA/2009/38 (H1N1) — Pandemic Live Attenuated Influenza Vaccine (PLAIV) Candidate Strain A/17/CA/2009/38 (H1N1)
  Other Names: GPO Flu Vaccine-01
  Arms: A/17/CA/2009/38 (H1N1)
Other: Placebo:Stabilizer — 5% sucrose
  Arms: Stabilizer

SUMMARY:
The purpose of this study is to evaluate safety and reactogenicity of Pandemic Live Attenuated Influenza Vaccine (PLAIV) manufactured by GPO, Thailand, and to evaluate humoral immune response of the above vaccine after intranasal application by using HAI test, micro neutralization assays.

DETAILED DESCRIPTION:
Part A: 24 volunteers will be enrolled and divided into 2 groups -12 volunteers in each of 2 groups receiving either 5.0-6.5 log 10 EID50 or 6.6-7.5 log10 EID50 respectively. 9 who will received vaccine vaccine strain and 3 who will received placebo.

Part B: Total 324 participants will randomized into 2 group using 3:1 ratio (300 vaccines:100 placebos). There are 3 stratified age groups: >12-18 years, >18-49 years and >49 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 9 - >49 years old
* Having Thai ID card or equivalent
* Are seronegative to the specific H1N1 influenza virus determined by antibody titer less than 1:10 by HAI test to the corresponding antigen
* Anti HIV - Negative
* All hematology & biochemistry within normal range
* Able to read and write and sign written informed consent

Exclusion Criteria:

* Known history of egg allergy
* Having had recently influenza infection confirmed as H1N1 (indeed all other types if Influenza and vaccination with seasonal vaccine will not interfere)
* History of bronchial asthma
* History of chronic lung diseases
* History of chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression
* Acute infectious and noninfectious diseases (within 2 weeks)
* Exacerbation of chronic diseases or cancer or HIV positives
* Anamnestic leukocytosis, hepatitis B and C positives
* The volunteers who have been taking immunoglobulin products or have had a blood transfusion during past three months before the beginning of the experiment
* Participation in other research study
* Pregnancy or plan to become pregnant for 60 days after enrollment or breast feeding
* Any concomitant medication with Aspirin

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2009-09; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Systemic reaction and local reaction (vital sign, temperature) | 11/2 year

SECONDARY OUTCOMES:
Humoral immune response | 11/2 year
  Peak immunogenicity blood specimen and nasal washing for accessing immune response IgA.
  Nasal swab on D2, D3, D5, D7 after immunization. Blood for ASC assay at D0 (baseline) and D7 after each dose of vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Punnee Pitisuttithum, MBBS,DTM&HDipGrad, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand